Official title: How Many Opiates Should be Prescribed for Pain in Patients

Undergoing Hip Arthroscopy? NCT number: NCT04169113 Document date: 17Feb2020

Collected data was analyzed with the primary outcome being the average number of tablets utilized between groups. Secondary outcome measurements analyzed the total number of pills remaining, number of days opioids were required, and post-operative NPRS scores. Patient baseline characteristics, known predictors of opioid abuse <sup>14</sup> and surgical information are reported as means ± standard deviation for continuous variables and percentages for categorical data. The aforementioned characteristics were compared using Student's t-tests, Pearson Chi Squared tests, and Fisher's Exact tests as appropriate. P < 0.05 (two-tailed) was considered significant. We then assessed for risk factors for increased opioid use after surgery by performing univariate and multivariate analyses, treating tablets used after surgery as a continuous variable. All independent variables with P<0.1 were included in the multivariate analysis. All statistical analyses were performed using SPSS (Version 23).